CLINICAL TRIAL: NCT03534024
Title: The Effects of Nanomicelles Curcumin on Glycemic Control, Serum Lipid Profile ,Blood Pressure and Anthropometric Measurements in Patients With Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, clinical professor, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 207
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nanomicielle curcumin (Active Comparator)
  Interventions: Dietary Supplement: nanomicielle curcumin
- plecebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: nanomicielle curcumin — Participants will be selected from those referring to endocrinology clinics of Shohadaye YaftAbad and Pars Hospital (Tehran, Iran) who meet the inclusion criteria. Each subject will give informed written consent to participate in the study. 10 cc fasting blood samples will be collected from each subject at baseline and at the end of trial. Anthropometric parameters will be measured.In order to control the confounding factors in patients, they will be randomly assigned to receive either nanomicelle curcumin or placebo. nanomcelle curcumin and placebo supplements will be provided from the Elixir Nano Sina Company the patients will advise not to change their lifestyle during the study.
  Arms: nanomicielle curcumin
Dietary Supplement: placebo — Participants will be selected from those referring to endocrinology clinics of Shohadaye YaftAbad and Pars Hospital (Tehran, Iran) who meet the inclusion criteria. Each subject will give informed written consent to participate in the study. 10 cc fasting blood samples will be collected from each subject at baseline and at the end of trial. Anthropometric parameters will be measured.In order to control the confounding factors in patients, they will be randomly assigned to receive either nanomcielle curcumin or placebo. nanomcelle curcumin and placebo supplements will be provided from the Elixir Nano Sina Company the patients will advise not to change their lifestyle during the study.
  Arms: plecebo

SUMMARY:
Metabolic syndrome is a condition which is recognized by abdominal obesity, dyslipidemia, hyperglycemia, and hypertension. Curcumin has beneficial effects such as antioxidant and anti-inflammatory effects. nanomcielle curcumin will be used in this study because of the low bioavailability , fast metabolism and low absorption of curcumin powder. Therefore, this study is planned to determine the effects of supplementation of nanomicelle curcumin on glycemic control, serum lipid profile ,blood pressure and anthropometric measurements in patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 25<body mass index >40
* waist circumference >102 cm in men or >88 cm in women
* Fasting blood glucose >100 mg/dL
* Triglycerides (TG) > 150 mg/dL
* High density lipoprotein cholesterol (HDL-C) <50 in women or <40 in men
* Systolic blood pressure (SBP) >130 mmHg and diastolic blood pressure (DBP) >85mmHg

Exclusion Criteria:

* insulin administration for diabetes control
* hypo- or hyperthyroidism,
* renal failure or other chronic diseases
* pregnancy and breastfeeding
* taking weight loss supplements and obeying unusual weight loss plans

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-08-30 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
hemoglobin A1c (HbA1c) | 12 weeks
serum glucose | 12weeks
serum insulin | 12weeks
homeostatic model assessment of insulin resistance(HOMA-IR) | 12weeks
homeostatic model assessment of beta cell(HOMA-B) | 12weeks
serum triglyceride (TG) | 12 weeks
serum total Cholesterol | 12 weeks
serum LDL-C | 12 weeks
serum HDL-C | 12 weeks
systolic blood pressure | 12 weeks
diastolic blood pressure | 12 weeks
serum curcumin | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Golbon Sohrab, Tehran, National Nutrition and Food Technology Research Institute, Iran